CLINICAL TRIAL: NCT00598325
Title: Phase 2 Single Center, Open-label Study to Assess Immunogenicity and Safety of 6 Doses of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX®)in Smokers
Brief Title: Antibody and Safety Study of 6 Doses of NicVAX in Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nabi-4513
Record Dates: First submitted 2008-01-09; First posted 2008-01-21 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Smoking
Keywords: Nicotine; Vaccine; Immunogenicity; Tobacco; Habits
MeSH Terms: conditions — Smoking; Habits | interventions — NicVAX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NicVAX (Experimental)
  Interventions: Biological: 3'-aminomethyl-Nic r-EPA Conjugate (NicVAX®)
- NicVAX Lot 2 (Experimental): 2nd cohort receives a different lot of vaccine from the 1st cohort
  Interventions: Biological: 3'-aminomethyl-Nic r-EPA Conjugate (NicVAX®)

INTERVENTIONS:
Biological: 3'-aminomethyl-Nic r-EPA Conjugate (NicVAX®) — 1.0 ml injection IM given every 4 weeks (weeks 0, 4, 8, 12, 16)
  Other Names: NicVAX

SUMMARY:
Prior clinical trials examined several schedules of a nicotine vaccine (NicVAX) for anti-nicotine antibody responses, and their impact on helping smokers quit. The best schedule so far has been one with doses at weeks 0, 4, 8, 16 and 26. This new study tests whether changing the schedule to weeks 0, 4, 8, 12 and 16 is an improvement for stimulating antibodies to nicotine. Routine vaccine safety information is also collected. Amendment 1 adds a 6th dose at week 26, and extends follow-up through week 52.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smoker, ≥10 cigarettes per day for 6 months, exhaled carbon monoxide ≥10 ppm
* Written informed consent
* Negative urine pregnancy test, and willing to use birth control during the study, if applicable

Exclusion Criteria:

* Prior exposure to nicotine vaccine
* Clinically significant allergic reactions, especially to components of the vaccine
* Serious or unstable clinical disease within the past 6 months
* Use of any smoking cessation therapy within 30 days preceding 1st dose
* Immunosuppression, due to: steroids or other immunosuppressants in the last 30 days, history of cancer or cancer treatment in the last 60 months, known HIV infection, or congenital or acquired immunodeficiency
* Use of any vaccine other than influenza vaccine within 30 days prior to each study dose
* Use of another IND drug or device within 30 days preceding 1st dose
* Inability to follow the protocol, or illicit drug use in the past 12 months, or psychiatric disorder in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Anti-nicotine antibody concentration | 12 time points between screening and week 20

SECONDARY OUTCOMES:
Vaccine reactogenicity | for 7 days after each dose
Adverse events | for 30 weeks after 1st dose (4 wk after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- Accelovance, Inc., Rockville, Maryland, United States

REFERENCES:
- [Derived] Fahim RE, Kessler PD, Fuller SA, Kalnik MW. Nicotine vaccines. CNS Neurol Disord Drug Targets. 2011 Dec;10(8):905-15. doi: 10.2174/187152711799219343. PMID 22229310
- [Derived] Hatsukami DK, Jorenby DE, Gonzales D, Rigotti NA, Glover ED, Oncken CA, Tashkin DP, Reus VI, Akhavain RC, Fahim RE, Kessler PD, Niknian M, Kalnik MW, Rennard SI. Immunogenicity and smoking-cessation outcomes for a novel nicotine immunotherapeutic. Clin Pharmacol Ther. 2011 Mar;89(3):392-9. doi: 10.1038/clpt.2010.317. Epub 2011 Jan 26. PMID 21270788